CLINICAL TRIAL: NCT02788851
Title: The Relative Efficacy of Aerobic Exercise in the Treatment of Adults With Attention Deficit Hyperactivity Disorder (ADHD) Versus Medication Only and the Combination of the Two: A Pilot Study
Brief Title: The Effectiveness of Aerobic Exercise in the Treatment of Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Lily Hechtman, Professor of Psychiatry and Pediatrics; Director of Research - Division of Child Psychiatry, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUHC-15-226
Record Dates: First submitted 2016-05-12; First posted 2016-06-02 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Stimulant Medication; Exercise; Functional Outcome; Effectiveness; Symptoms
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Activity | interventions — Guanfacine; Methylphenidate; Dextroamphetamine; SLI381; Lisdexamfetamine Dimesylate; Atomoxetine Hydrochloride; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Medication only (Active Comparator): Stimulant or non-stimulant medication only - Methylphenidate compounds and /or Amphetamine compounds and/or Strattera or Guanfacine. Investigators will be using a product approved for clinical use in Canada), with dose optimized for each participant based on report of efficacy and side effects. Once on an optimal dose of stimulant or non-stimulant medication they will attend 8 weekly education sessions about ADHD.
  Interventions: Drug: Methylphenidate compounds and /or Amphetamine compounds and/or Strattera or Guanfacine
- Aerobic Exercise only (Experimental): Participants attend a structured aerobic exercise class, twice a week for 8 weeks.
  Interventions: Behavioral: Aerobic Exercise
- Combination Group (Active Comparator): Participants assigned to this group will be optimally medicated (either stimulant or non-stimulant medication - approved for clinical use in Canada) and will attend a structured aerobic exercise class, twice a week for 8 weeks.
  Interventions: Drug: Methylphenidate compounds and /or Amphetamine compounds and/or Strattera or Guanfacine; Behavioral: Aerobic Exercise

INTERVENTIONS:
Drug: Methylphenidate compounds and /or Amphetamine compounds and/or Strattera or Guanfacine — Medication is titrated over a 4-week period with stepwise increments each week. Participants and their significant others will complete ADHD symptom scales at baseline and before each medication visit. Participants also complete a side effects scale at baseline and before each medication visit. The gradual increase will continue until there is no further improvement in symptoms and in the Clinical Global Improvement Scale or side effects are such that further increases are not indicated. Once the optimal dose is reached, the participant will remain on this dose for the remainder of the study. Additionally, once the optimal dose is reached participants will attend 8 weekly educational sessions about ADHD in adulthood.
  Other Names: Ritalin; Concerta; Biphentin; Dexedrine; Adderall XR; Vyvanse; Strattera; Guanfacine; Intuniv
  Arms: Combination Group; Medication only
Behavioral: Aerobic Exercise — Participants will attend a structured aerobic exercise class twice a week for 8 weeks. Each class will last 60 minutes.
  Arms: Aerobic Exercise only; Combination Group

SUMMARY:
The purpose of this project is to evaluate the effectiveness of a structured aerobic exercise intervention for adults with Attention-Deficit/Hyperactivity Disorder (ADHD) with and without medication and compare it to medication alone. Participants will be randomly assigned to medication only + education, aerobic exercise intervention only, and combined aerobic exercise and medication groups. Participants will be evaluated at baseline, following medication optimization (for medicated groups), following 8 weeks of intervention, after 3 months of follow-up, and after 6 months of follow-up. The investigators hypothesize that the combined group will have the best outcome at all evaluation points and that treatment gains will be maintained throughout the follow-up period if the assigned treatments are continued.

DETAILED DESCRIPTION:
Background: Several interventional studies have shown improvement in core symptoms of Attention-Deficit Hyperactivity Disorder (ADHD) with aerobic exercise as an add-on therapy for children with ADHD treated with stimulants. Studies in the general population have shown that aerobic exercise in adults may improve cognitive function in general and executive function in particular. Although non-medication treatment for ADHD has focused on cognitive training in addition to medication, some evidence indicate that intense aerobic exercise impacts brain structure, improves brain function, and has effects similar to stimulant medication.

Objectives: To assess the effectiveness, regarding ADHD symptoms, of an eight week aerobic exercise intervention, medication, and the combination of both aerobic exercise and medication treatments for adults with ADHD. The secondary objectives are to determine the effectiveness of these treatments on social skills, as measured by functioning in work, social, and family situations; anxiety symptoms; depressive symptoms; self-esteem; and the effect of motivation for exercise on adherence to exercise treatment.

Hypothesis: Investigators hypothesize that the combined group which receives aerobic exercise and medication intervention will have the greatest improvement in both primary and secondary outcome measures; that treatment gains will be maintained at follow-up only if treatments are continued.

Methods: Participants will be randomly assigned to one of three groups:

1. Aerobic exercise intervention only. Participants of this group will meet twice a week for 8 consecutive weeks. Each meeting will involve 1 hour of moderate-vigorous intensity aerobic exercise.
2. Medication treatment only. Participants of this group will receive optimal medication for them and will gradually be titrated up to their optimal dose. Once they are optimally titrated, they will attend 8 weekly sessions of an education class, which will focus on different topics of adult ADHD. These meetings will last 1 hour each week. Educational meetings are meant to control for group effects of the exercise group intervention.
3. Medication combined with aerobic-exercise intervention. Participants of this group will receive optimal medication for them and will gradually be titrated up to their optimal dose. When the participants of this group will be at their optimal medication dose, they will begin the aerobic exercise classes twice a week for 8 weeks. They will not receive the educational sessions.

Randomization will be stratified by sex, age and the degree of physical activity per week. Power analyses indicate that 23 participants are needed per each treatment arm, accounting for a dropout rate of 20%. Therefore initial enrollments should be at minimum 69 patients for all three arms, at least 23 patients per arm. There will 2 groups in each arm of the study, accounting for 10-15 participants per group at any one time.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for adult ADHD of any of three presentations (inattentive, hyperactive impulsive, combined) via Conners Adult ADHD Diagnostic Interview for the DSM-5 (CAARD-D) and clinician's assessment;
2. Barkley Childhood and Current Symptom of ADHD (1998) completed by self and informants (parents or siblings for childhood symptoms, spouses or co-workers for current symptoms). Required cut off on these scales are scores 1.5 Standard Deviation above relevant gender and age norms;
3. Conners Adult ADHD Rating Scale (1999) completed by self and informants, such as spouses or co-workers for current ADHD symptoms. Required cut off on these scales are scores 1.5 Standard Deviation above relevant gender and age norms;
4. Between 18 and 60 years old
5. Be able to give informed consent and comply with study procedures;
6. I.Q. of 85 or above on Wechsler Adult Intelligence Scale - Third Edition (WAIS-III) by three verbal and three nonverbal subtests
7. Adequate command of English to be able to participate in the group treatment.
8. Written permission from a family physician to participate in aerobic exercise and no contra-indications for stimulant medication.

Exclusion Criteria:

1. Psychotic symptoms, past or current;
2. Current psychiatric comorbidity, which needs ongoing medication treatment e.g. bipolar disorder, major depression, suicidality, anxiety, current substance use disorder (must be free of substance abuse for 12 months);
3. Medical condition that preclude use of the stimulant medication, e.g. hypertension, cardiac disease, Tourette syndrome, etc.
4. Organic mental disorders or other significant neurological disorders, e.g. epilepsy, head injury, chorea, multiple sclerosis.
5. Pregnant or breastfeeding women.
6. Patients currently involved in intensive aerobic exercise, two hours per week or more.
7. Patients who are currently effectively treated for ADHD.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported ADHD symptoms (measured via Barkley's Current ADHD Symptoms Scale) - Change from baseline | At baseline; once optimally titrated (about 5 weeks to reach this dose for medication groups); after 8 weeks of intervention (aerobic exercise or educational sessions); 3 months after the end of intervention; 6 months after the end of intervention

SECONDARY OUTCOMES:
Depression symptoms (via the Beck Depression Inventory) - Change from baseline | At baseline; once optimally titrated (about 5 weeks to reach this dose for medication groups); after 8 weeks of intervention (aerobic exercise or educational sessions); 3 months after the end of intervention; 6 months after the end of intervention
Anxiety Symptoms (measured via the Beck Anxiety Inventory) - Change from baseline | At baseline; once optimally titrated (about 5 weeks to reach this dose for medication groups); after 8 weeks of intervention (aerobic exercise or educational sessions); 3 months after the end of intervention; 6 months after the end of intervention
Global functional impairment (measured via the Sheehan Disability Scale) - Change from baseline | At baseline; once optimally titrated (about 5 weeks to reach this dose for medication groups); after 8 weeks of intervention (aerobic exercise or educational sessions); 3 months after the end of intervention; 6 months after the end of intervention
Self-esteem (measured via the Index of Self-Esteem) - Change from baseline | At baseline; once optimally titrated (about 5 weeks to reach this dose for medication groups); after 8 weeks of intervention (aerobic exercise or educational sessions); 3 months after the end of intervention; 6 months after the end of intervention
Dyadic adjustment (for those married or cohabiting, measured via the Dyadic Adjustment Scale) - Change from baseline | At baseline; once optimally titrated (about 5 weeks to reach this dose for medication groups); after 8 weeks of intervention (aerobic exercise or educational sessions); 3 months after the end of intervention; 6 months after the end of intervention
Motivation to exercise (measured via the Physical Activity and Leisure Motivation Scale) - Change from baseline | At baseline; once optimally titrated (about 5 weeks to reach this dose for medication groups); after 8 weeks of intervention (aerobic exercise or educational sessions); 3 months after the end of intervention; 6 months after the end of intervention
Stimulant medication side effects (measured via the Canadian ADHD Resource Alliance (CADDRA) Patient ADHD Medication Form) | Completed before each medication visit, every 1 - 2 weeks up to 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Lily Hechtman, MD, FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis CL, Tomporowski PD, McDowell JE, Austin BP, Miller PH, Yanasak NE, Allison JD, Naglieri JA. Exercise improves executive function and achievement and alters brain activation in overweight children: a randomized, controlled trial. Health Psychol. 2011 Jan;30(1):91-8. doi: 10.1037/a0021766. PMID 21299297
- [Background] Kang KD, Choi JW, Kang SG, Han DH. Sports therapy for attention, cognitions and sociality. Int J Sports Med. 2011 Dec;32(12):953-9. doi: 10.1055/s-0031-1283175. Epub 2011 Nov 8. PMID 22068930
- [Background] Smith AL, Hoza B, Linnea K, McQuade JD, Tomb M, Vaughn AJ, Shoulberg EK, Hook H. Pilot physical activity intervention reduces severity of ADHD symptoms in young children. J Atten Disord. 2013 Jan;17(1):70-82. doi: 10.1177/1087054711417395. Epub 2011 Aug 25. PMID 21868587
- [Background] Tantillo M, Kesick CM, Hynd GW, Dishman RK. The effects of exercise on children with attention-deficit hyperactivity disorder. Med Sci Sports Exerc. 2002 Feb;34(2):203-12. doi: 10.1097/00005768-200202000-00004. PMID 11828226
- [Background] Kramer AF, Hahn S, Cohen NJ, Banich MT, McAuley E, Harrison CR, Chason J, Vakil E, Bardell L, Boileau RA, Colcombe A. Ageing, fitness and neurocognitive function. Nature. 1999 Jul 29;400(6743):418-9. doi: 10.1038/22682. No abstract available. PMID 10440369
- [Background] Fiatarone Singh MA, Gates N, Saigal N, Wilson GC, Meiklejohn J, Brodaty H, Wen W, Singh N, Baune BT, Suo C, Baker MK, Foroughi N, Wang Y, Sachdev PS, Valenzuela M. The Study of Mental and Resistance Training (SMART) study-resistance training and/or cognitive training in mild cognitive impairment: a randomized, double-blind, double-sham controlled trial. J Am Med Dir Assoc. 2014 Dec;15(12):873-80. doi: 10.1016/j.jamda.2014.09.010. Epub 2014 Oct 23. PMID 25444575
- [Background] Verret C, Guay MC, Berthiaume C, Gardiner P, Beliveau L. A physical activity program improves behavior and cognitive functions in children with ADHD: an exploratory study. J Atten Disord. 2012 Jan;16(1):71-80. doi: 10.1177/1087054710379735. Epub 2010 Sep 13. PMID 20837978
- [Background] Robinson AM, Bucci DJ. Individual and combined effects of physical exercise and methylphenidate on orienting behavior and social interaction in spontaneously hypertensive rats. Behav Neurosci. 2014 Dec;128(6):703-12. doi: 10.1037/bne0000015. Epub 2014 Aug 25. PMID 25150541
- [Background] Freeman MP. ADHD and pregnancy. Am J Psychiatry. 2014 Jul;171(7):723-8. doi: 10.1176/appi.ajp.2013.13050680. PMID 24980168
- [Background] Cole CR, Blackstone EH, Pashkow FJ, Snader CE, Lauer MS. Heart-rate recovery immediately after exercise as a predictor of mortality. N Engl J Med. 1999 Oct 28;341(18):1351-7. doi: 10.1056/NEJM199910283411804. PMID 10536127
- [Background] Nishime EO, Cole CR, Blackstone EH, Pashkow FJ, Lauer MS. Heart rate recovery and treadmill exercise score as predictors of mortality in patients referred for exercise ECG. JAMA. 2000 Sep 20;284(11):1392-8. doi: 10.1001/jama.284.11.1392. PMID 10989401
- [Background] Gajria K, Lu M, Sikirica V, Greven P, Zhong Y, Qin P, Xie J. Adherence, persistence, and medication discontinuation in patients with attention-deficit/hyperactivity disorder - a systematic literature review. Neuropsychiatr Dis Treat. 2014 Aug 22;10:1543-69. doi: 10.2147/NDT.S65721. eCollection 2014. PMID 25187718
- [Background] Joseph A, Cloutier M, Guerin A, Nitulescu R, Sikirica V. Treatment outcomes after methylphenidate in adults with attention-deficit/hyperactivity disorder treated with lisdexamfetamine dimesylate or atomoxetine. Patient Prefer Adherence. 2016 Mar 24;10:391-405. doi: 10.2147/PPA.S98498. eCollection 2016. PMID 27069357
- [Background] Barnes DE, Santos-Modesitt W, Poelke G, Kramer AF, Castro C, Middleton LE, Yaffe K. The Mental Activity and eXercise (MAX) trial: a randomized controlled trial to enhance cognitive function in older adults. JAMA Intern Med. 2013 May 13;173(9):797-804. doi: 10.1001/jamainternmed.2013.189. PMID 23545598
- [Background] Safren SA, Sprich S, Mimiaga MJ, Surman C, Knouse L, Groves M, Otto MW. Cognitive behavioral therapy vs relaxation with educational support for medication-treated adults with ADHD and persistent symptoms: a randomized controlled trial. JAMA. 2010 Aug 25;304(8):875-80. doi: 10.1001/jama.2010.1192. PMID 20736471